CLINICAL TRIAL: NCT06807450
Title: Repair of Oronasal Fistula Using Interpositional Buccal Pad of Fat as a Free Graft in a Cleft Palate Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, mona samy sheta, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202014
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cleft Palate
Keywords: oro-nasal fistula; cleft palate; buccal pad of fat free graft
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repair of oro-nasal fistula using two layers (Experimental): the fistula will be closed using two layers nasal layer by turning over the fistula margin and closure with 4/0 vicryl oral layer using two flap palatoplasty with relaxing incision around the alveolar margin and approximate at the midline using 4/0 vicryl
  Interventions: Procedure: closure of oro-nasal fistula in cleft palate patients
- repair of oro-nasal fistula using two layers with interpositional buccal pad of fat free graft (Experimental): the fistula will be closed using two layers nasal layer by turning over the fistula margin and closure with 4/0 vicryl oral layer using two flap palatoplasty with relaxing incision around the alveolar margin and approximate at the midline using 4/0 vicryl then a free graft of buccal pad of fat will be obtained and inserted between the two layers
  Interventions: Procedure: closure of oro-nasal fistula in cleft palate patients

INTERVENTIONS:
Procedure: closure of oro-nasal fistula in cleft palate patients — group I : Oro-nasal fistula will be closed in two layers, nasal layer by closing the fistula margin and turning over of flap and oral layer will be closed using two flap palatoplasty group II; the same procedure with insertion of free graft of buccal pad of fat between oral and nasal layers
  Other Names: repair of oro-nasal fistula in cleft palate patients

SUMMARY:
36 cleft palate patients had residual oronasal fistula included in this study divided randomly to two groups group I (control group): the fistula was repaired using two layers (oral and nasal layers) group II (study group): The fistula was repaired using two layers (oral and nasal layers ) with interpositional free buccal pad of fat graft between two layers

DETAILED DESCRIPTION:
36 cleft palate patients had residual oronasal fistula included in this study devided randomly to two groups group I (control group):the fistula was repaired using two layers nasal layer:closed by turn-in flaps, taken from around the margins of the fistula by making incision around margins of distance slightly larger than half of diameter of fistula bilaterally, then closed by inverted interrupted suture Vicry l 4/0.

oral layer:(Bardach two-flap palatoplasty) was used and raised on opposite sides of the cleft palate and brought together in the midline to create a continuous palate

group II (study group): The fistula was repaired using two layers (oral and nasal layers ) as group I with buccal pad of fat free graft was taken through veastibular incision at zygomatic buttress then blunt dissection to get buccal fat which was released from its pedicle and inserted between oral and nasal layers.

ELIGIBILITY:
Inclusion Criteria:

* cleft palate patients with oro-nasal fistula fistula in hard palate

Exclusion Criteria:

* syndromatic patients

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
evaluation of wound healing | one month
  five level
  1. very poor
  2. poor
  3. good
  4. very good
  5. excellent
recurrence of oro-nasal fistula | one -3 months
  present or abscent

SECONDARY OUTCOMES:
postoperative pain | one month
  using visual analogue scale (0-10) 0: no pain 10: the worest pain

CONTACTS AND LOCATIONS:
Overall Officials: mona s sheta, lecturer, Principal Investigator — Tanta University
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt